CLINICAL TRIAL: NCT01306461
Title: A Phase III, Randomized, Double-masked 6-month Trial to Compare the Efficacy and Safety of the Preservative-free Fixed-dose Combination of Tafluprost and Timolol Eye Drops to Those of Tafluprost and Timolol Eye Drops Given Concomitantly in Patients With Open Angle Glaucoma or Ocular Hypertension
Brief Title: Tafluprost-Timolol Fixed Dose Combination Non-Inferiority Study Against Concomitant Administrations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Oy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201051
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Ocular Hypertension; Open-angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — Timolol; tafluprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Timolol and Tafluprost (Active Comparator): Concomitant administration of preservative-free timolol and tafluprost eye drops
  Interventions: Drug: Timolol and Tafluprost
- Fixed Dose Combination of tafluprost and timolol (Experimental): Preservative-free Fixed Dose Combination of tafluprost and timolol eye drops
  Interventions: Drug: Fixed Dose Combination of tafluprost and timolol

INTERVENTIONS:
Drug: Timolol and Tafluprost — Preservative-free Timolol eye drops administered twice daily concomitantly with preservative-free Tafluprost eye drops administered once daily
  Treatment period 6 months
  Arms: Timolol and Tafluprost
Drug: Fixed Dose Combination of tafluprost and timolol — Preservative-free Fixed Dose Combination of tafluprost and timolol eye drops administered once daily.
  For masking purposes also: vehicle for timolol administered twice daily
  Treatment period 6 months
  Arms: Fixed Dose Combination of tafluprost and timolol

SUMMARY:
The purpose of this study is to compare the efficacy and safety of the preservative-free fixed-dose combination of tafluprost and timolol (FDC) to concomitant administration of tafluprost and timolol.

This study will enroll patients who have ocular hypertension or glaucoma.

The study schedule includes seven visits to the study site and three stages:

* washout of 5 days to 4 weeks depending on current glaucoma medication (if any)
* 6-month study treatment period
* 1-3 weeks post-study period

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more
* A diagnosis of ocular hypertension or open-angle glaucoma
* Meet specific IOP level at visit 1 (screening)and visit 2 (baseline)
* Meet specific visual acuity score
* Are willing to follow instructions
* Have provided a written informed consent

Exclusion Criteria:

* Females who are pregnant, nursing or planning pregnancy
* IOP greater than 36 mmHg at any time point at screening or baseline
* Diagnosis of angle-closure glaucoma or secondary glaucoma other than capsular or pigmentary glaucoma in either eye
* Suspected contraindication or hypersensitivity to study medications tafluprost or timolol (e.g. asthma, low pulse) or to wash-out medication brinzolamide
* Glaucoma filtration surgery or any other ocular surgery (including ocular laser procedures) within 6 months prior to Screening
* Use of contact lenses at Screening or during the study
* Presence of any abnormality or significant illness that could be expected to interfere with the patient safety or study parameters
* Current participation in another clinical trial within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the average diurnal intra-ocular pressure (IOP) at 6 months | 6 months

SECONDARY OUTCOMES:
Change from baseline in average diurnal IOP at 2 weeks, 6 weeks and 3 months | 2 weeks, 6 weeks and 3 months
Change from baseline in timewise IOPs | 2 weeks, 6 weeks, 3 months and 6 months
  Change from baseline in timewise IOPs (at 8:00, 10:00, 16:00) at 2 weeks, 6 weeks, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Auli Ropo, M.D., Study Director — Santen Oy; Clemens Vass, M.D., Principal Investigator — Medical University Vienna, Austria; Marieta Kostianeva, M.D., Principal Investigator — University Mulitiprofile Hospital for Active Treatment Sv.Georgi, Bulgaria; Eva Ruzickova, M.D., Principal Investigator — Vseobecna fakultni nemocnice v Praze, Czech Republic; Gábor Holló, Principal Investigator — Semmelweis Egyetem, Hungary; Guna Laganovska, M.D., Principal Investigator — P. Stradina Clinical University Hospital, Latvia; Maria L. Ribeiro, M.D., Principal Investigator — Aibili-Associação p/ Investigação Biomédica e Inovação em Luz e Imagem (AIBILI), Portugal; Julián García-Feijóo, M.D., Principal Investigator — Hospital Clinico San Carlos, Spain
Locations (1):
- Debrecen, Hungary